CLINICAL TRIAL: NCT01531322
Title: A Phase 1 Open-label Study to Assess the Safety and Tolerability of a Single Dose of 13-valent Pneumococcal Conjugate Vaccine in Healthy Chinese Adults, Children and Infants
Brief Title: A Study Assessing 13-valent Pneumococcal Conjugate Vaccine in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B1851046; 6096A1-1000
Record Dates: First submitted 2011-08-12; First posted 2012-02-10 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Pneumococcal Infection
Keywords: 13vPnC; Healthy subjects; China
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Adults aged 18 through 55 years (before the fifty sixth birthday)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- Group 2 (Experimental): Children aged 3 through 5 years (before the sixth birthday)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- Group 3 (Experimental): Infants aged approximately 2 months (42 to 98 days)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — suspension in prefilled syringe for intramuscular injection, 0.5 mL, only one dose
  Arms: Group 1
Biological: 13-valent Pneumococcal Conjugate Vaccine — suspension in prefilled syringe for intramuscular injection, 0.5 mL, only one dose
  Arms: Group 2
Biological: 13-valent Pneumococcal Conjugate Vaccine — suspension in prefilled syringe for intramuscular injection, 0.5 mL, only one dose
  Arms: Group 3

SUMMARY:
This study will assess the safety and tolerability of a single dose of 13-valent Pneumococcal Conjugate Vaccine for approximately 1 month after vaccination sequentially in healthy Chinese adults aged 18 through 55 years, followed by children aged 3 through 5 years, and then infants aged approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of enrollment is:

   * 18 through 55 years (before the fifty sixth birthday) for Group 1.
   * 3 through 5 years (before the sixth birthday) for Group 2.
   * 42 to 98 days for Group 3.
2. Healthy subject as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal vaccine.
* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with pneumococcal vaccine.

Ages: 42 Days to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting Adverse Events | Baseline to Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Pfizer Investigational Site, Huaian, Jiangsu
  - Pfizer Investigational Site, Nanjing, Jiangsu

REFERENCES:
- [Derived] Zhu F, Hu Y, Liang Q, Young M Jr, Zhou X, Chen Z, Liang JZ, Gruber WC, Scott DA. Safety and tolerability of 13-valent pneumococcal conjugate vaccine in healthy Chinese adults, children and infants. Ther Adv Drug Saf. 2015 Dec;6(6):206-11. doi: 10.1177/2042098615613985. PMID 26668712
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851046&StudyName=A%20Study%20Assessing%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20in%20Healthy%20Chinese%20Subjects